CLINICAL TRIAL: NCT05710783
Title: Phase II/III Parallel, Double-blind, Non-inferiority Study With Active Control, to Evaluate the Immunogenicity and Safety of a Booster Immunization Scheme With a Single Intramuscular Dose of the Recombinant Vaccine Against SARS-CoV-2
Brief Title: Phase II/III Study of the AVX/COVID-12 Vaccine Against COVID-19 Applied as a Booster.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Laboratorio Avi-Mex, S.A. de C.V. (Industry)
Collaborators: National Council of Science and Technology, Mexico (Other); Instituto Nacional de Enfermedades Respiratorias (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AVX-SARS-CoV-2-VAC-005
Record Dates: First submitted 2022-12-21; First posted 2023-02-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: SARS-CoV-2 Infection
Keywords: Newcastle Disease Virus; rNDV; COVID-19; SARS-Cov-2 Vaccine; Booster COVID-19 Vaccine
MeSH Terms: conditions — COVID-19 | interventions — ChAdOx1 nCoV-19

STUDY DESIGN:
Intervention Model Description: Immuno-bridging
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization of patients shall be carried out by a computerized system. Once the informed consent signed, the patient shall be allocated with a number coding with all his/her pseudonymously information during collection and completely anonymised during analysis.
  The randomization of the first 400 study subjects will include, in addition to 1:1 randomization (experimental vaccine: active control), randomization to participate as a subsample subject for cellular immune response determinations.
  Once the 1664 subjects have been randomised, the following study subjects shall be designated as experimental vaccine receptors until have enrolled all the study subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Phase II - Experimental (Experimental): AVX-COVID/12 Dose: 10^8.0 EID50/ intramuscular dose Study parameters: Safety, Serological response, Cellular response
  Interventions: Biological: AVX-COVID/12
- Phase II - Active Control (Active Comparator): ChAdOx-1-S[recombinant]) intramuscular Study parameters: Safety, Serological response, Cellular response
  Interventions: Biological: ChAdOx-1-S[recombinant]
- Phase III - Experimental (Experimental): AVX-COVID/12 Intramuscular Dose: 10^8.0 EID50/ intramuscular dose Study parameters: Safety, Serological response
  Interventions: Biological: AVX-COVID/12
- Phase III - Active Control (Active Comparator): ChAdOx-1-S[recombinant]) intramuscular Study parameters: Safety, Serological response
  Interventions: Biological: ChAdOx-1-S[recombinant]
- Phase III - Security (Experimental): AVX-COVID/12 Intramuscular Dose: 10^8.0 EID50/ intramuscular dose Study parameters: Safety.
  Interventions: Biological: AVX-COVID/12
- Phase II- Experimental (Experimental): AVX-COVID/12 Dose: 10^8.0 EID50/ intramuscular dose Study parameters: Safety, Serological response.
  Interventions: Biological: AVX-COVID/12
- Phase II- Active Control (Active Comparator): ChAdOx-1-S[recombinant]) intramuscular Study parameters: Safety, Serological response.

INTERVENTIONS:
Biological: AVX-COVID/12 — Single dose IM administration of a Recombinant Newcastle Disease Virus Vectored Vaccine for SARS-CoV-2
  Other Names: Recombinant NDV Vectored Vaccine for SARS-CoV-2
  Arms: Phase II - Experimental; Phase II- Experimental; Phase III - Experimental; Phase III - Security
Biological: ChAdOx-1-S[recombinant] — Single dose IM administration of ChAdOx1 nCOV-19 (Astra-Zeneca) adenovirus-vectored vaccine
  Other Names: AstraZeneca COVID vaccine
  Arms: Phase II - Active Control; Phase III - Active Control

SUMMARY:
This is a phase II/III parallel, double-blind, active-controlled, non-inferiority study to evaluate immunogenicity and safety of a booster immunization scheme of a single intramuscular dose of the recombinant vaccine against SARS-CoV-2 (AVX/COVID-12 vaccine) based on live recombinant Newcastle disease virus (rNDV) vector in healthy adults with a history of vaccination against COVID-19. The study is divided into two phases with immuno-bridging and 3000 healthy subjects showing evidence of prior immunity to SARS-CoV-2 are estimated to enrol. To verify non-inferiority in a determined number of subjects an intramuscular dose of the COVID-19 vaccine (ChAdOx-1-S[recombinant]) shall be used as active control in originally randomised subjects. The study shall be carried out in several sites of clinical research in Mexico.

DETAILED DESCRIPTION:
General objective:

To demonstrate immunogenicity and safety of the AVX/COVID-12 vaccine (108.0 EID50/dose) as a single intramuscular booster shot in previously vaccinated subjects and prove non-inferiority producing neutralizing antibodies anti-COVID-19 from 14 days after administration in comparison to the active control, whose efficacy has been formerly established in a placebo-controlled clinical study.

Primary objective:

Phase II:

To demonstrate immunogenicity of the AVX/COVID-12 vaccine (108.0 EID50/dose) as a single intramuscular booster shot to increase levels of Spike protein to ACE2 binding-inhibitory antibodies, as well as to increase titres of neutralizing antibodies anti-COVID-19 from 14 days after vaccine administration.

Phase III:

To demonstrate non-inferiority of the AVX/COVID-12 vaccine (108.0 EID50/dose) as a single intramuscular booster shot for seroconversion and production of neutralizing antibodies anti-COVID-19 from 14 days after vaccine administration compared to active control, whose efficacy has been formerly established in a placebo-controlled clinical study.

Secondary objectives:

Phase II:

To evaluate the extent of the increase in the neutralizing titres after 0, 14, 90 and 180 days of administration of the AVX/COVID-12 vaccine (108.0 EID50/dose) as a single intramuscular booster shot.

To evaluate production of interferon-gamma by peripheral blood T lymphocytes in response to the Spike protein or its derivatives peptides stimulation following 0, 14, 90 and 180 days of administration of the AVX/COVID-12 vaccine (108.0 EID50/dose) as a single intramuscular booster shot in a subgroup of subjects randomly selected among the study population.

To compare production of interferon-gamma by peripheral blood T lymphocytes in response to the Spike protein or its derivatives peptides stimulation following 0, 14, 90 and 180 days of administration of the AVX/COVID-12 vaccine (108.0 EID50/dose) as a single intramuscular booster shot in a subgroup of subjects randomly selected among the study population to production in subjects vaccinated with active control.

Phase III:

To document the incidence of symptomatic COVID-19 disease cases in both groups (experimental vaccine and active control) from 14 days after administration.

To document the incidence of severe or mortality COVID-19 disease cases in both groups (experimental vaccine and active control) from 14 days after administration.

Safety objective (primary):

Both Phases:

To evaluate safety of AVX/COVID-12 vaccine immunization as a single intramuscular booster shot in comparison to the active control.

Exploratory objectives:

Phase II:

To evaluate the extent of the increase in following neutralizing titres 0, 14, 90 and 180 days of administration of the AVX/COVID-12 vaccine (108.0 EID50/dose) as a single intramuscular booster shot as per the history of immunization/infection at the time of enrolment.

To evaluate the neutralizing capacity of anti-SARS-CoV-2 antibodies gained following 0, 14, 90 and 180 days of administration of the AVX/COVID-12 vaccine (108.0 EID50/dose) as a single intramuscular booster shot in neutralization tests of pseudovirus expressing Spike proteins derived from SARS-CoV-2 variants of concern.

To evaluate production of cytokines by peripheral blood T lymphocytes in response to the Spike protein or its derivatives (peptides) stimulation following 0, 14, 90 and 180 days of administration of the AVX/COVID-12 vaccine (108.0 EID50/dose) as a single intramuscular booster shot in a subgroup of subjects randomly selected among the population study.

To compare production of cytokines by peripheral blood T lymphocytes in response to the Spike protein or its derivatives (peptides) stimulation following 0, 14, 90 and 180 days of administration of the AVX/COVID-12 vaccine (108.0 EID50/dose) as a single intramuscular booster shot in a subgroup of subjects randomly selected among the population study to production in subjects vaccinated with active control.

Phase III:

To compare geometric means of neutralizing titres after AVX/COVID-12 (108.0 EID50/dose) vaccination as a single intramuscular booster shot in the following active-controlled subgroups:

* Subjects younger than 65 years.
* Subjects older than 65 years.
* Subjects with at least one comorbidity (any).
* Subjects with obesity (BMI >30).
* Subjects with Diabetes Mellitus.
* Subjects with hypertension.
* Subjects with smoking history.
* Subjects with asthma.
* Subjects with cardiovascular disease.
* Subjects with chronic obstructive pulmonary disease.
* Subjects with chronic renal disease.
* Subjects with liver disease.
* Subjects with cancer history.

Clinical trial hypothesis:

Phase II:

In subjects with prior anti-SARS-CoV-2 vaccination longer than 4 months ago, 14 days after intramuscular administration of the AVX/COVID-12 vaccine, ≥80% of the subjects showed an inhibitory capacity of the receptor-binding domain (spike protein binds to ACE2) above 95% and levels of neutralizing titres statistically greater than baseline tires (vaccination day).

Phase III:

Immunogenicity assessed as seroconversion rate and production of neutralizing antibodies after administration of the AVX/COVID-12 vaccine as a single intramuscular booster shot of 108.0 EID50/dose showed non-inferiority to active control from 14 days after administration.

Justification of the product use in clinical research.

Nonclinical studies and Phase I clinical study have shown safety of the AVX/COVID-12 vaccine by intramuscular route. Signs of immunogenicity in several animals are clear. Evaluation of the immune response in healthy volunteers in the Phase I clinical study after administration of the vaccine by intramuscular route as a single dose of 108.0 EID50/dose showed immunogenicity of the vaccine. Partial reports from a Phase II boosting study in subjects with low levels of immunity at the time of enrolment strongly suggest the vaccine is safe and immunogenic in this population. Altogether, these data justify the continuation of the AVX/COVID-12 vaccine development program. Due to the advanced stage of the pandemics and vaccination programs worldwide, it is important to assess the capacity of the AVX/COVID-12 vaccine to boost the pre-existing immunity in open previously vaccinated population.

Study design:

A phase II/III parallel, double-blind, active-controlled, non-inferiority study to evaluate immunogenicity and safety of a booster immunization scheme with a single intramuscular dose of the recombinant vaccine against SARS-CoV-2 (AVX/COVID-12 vaccine) based on live recombinant Newcastle disease virus (rNDV) vector in healthy adults with a history of vaccination against COVID-19.

Summarised description of Phase II design:

Subjects who meet the study inclusion and not exclusion criteria shall be randomised (1:1) to receive the AVX/COVID-12 vaccine or active control.

From the first 400 subjects of study samples corresponding to the efficacy criteria for Phases II and III shall be collected (including samples to determine cell response in a randomly-defined subgroup).

If at the end of the main endpoint assessment of the study phase corresponding to Phase II (day 14) it is determined the intervention with AVX-COVID-12 vaccine did not meet the specified objective (i. e., neutralizing capacity above 95% was not showed in 80% of the population vaccinated in surrogate testing and a significant change when comparing the geometric means of population neutralizing antibodies titres from days 0 to 14) the enrolment shall be stopped in order to meet the criteria related to the Phase III objectives, otherwise the enrolment shall continue consecutively.

Additionally, the first 400 subjects enrolled (corresponding to Phase II (200 vaccinated with the experimental vaccine and 200 with the active control)) shall be evaluated 90 and 180 days after vaccination to determine the humoral immune response performance at these moments.

A sub-sample of 100 subjects randomly selected (50 experimental vaccine and 50 active control) shall be evaluated regarding cell-mediated immune response in addition to the humoral response at the time of enrolment and 14, 90 and 180 days after vaccination.

Comparison of the safety evaluation related to Phase II shall be carried out with the population receiving active control as reference.

An interim futility analysis shall be carried out for non-inferiority criteria of Phase III at the end of enrolment corresponding to Phase II by Fleming-alpha spending function.

Summarised description of Phase III design:

In total 3832 subjects shall be enrolled divided into 3000 subjects to receive the experimental vaccine (2168 + 832 (632 Phase III + 200 from Phase II/III)) and 832 subjects (632 Phase II + 200 from Phase II/III) will receive active control.

The first 1664 subjects enrolled shall be randomised 1:1 to receive the experimental vaccine or active control and at the end of this phase the subsequent number of subjects enrolled shall receive only the experimental vaccine up to 3000 subjects.

From the first 1664 subjects of study (832 randomised to receive the experimental vaccine and 832 vaccinated with active control) samples shall be collected on days 0 and 14 to determine total titres of anti-S IgG, total titres of anti-N IgG and anti-SARS-CoV-2 neutralizing titres.

Three thousand subjects from safety population and 832 subjects vaccinated with active control shall be followed-up to 180 days to detect symptomatic cases of COVID-19 proved with genetic material detection from nasal/mouth mucus by PCR.

ELIGIBILITY:
Inclusion Criteria:

1. People ≥18 years old.
2. Any genre.
3. Have received their informed consent.
4. Negative PCR test for SARS-CoV-2 during the screening visit.
5. Negative pregnancy test in women with child-bearing potential.
6. Commitment to maintain adequate prevention measures to avoid contagion by SARS-CoV-2 throughout their participation in the study considering their strict following for the first 14 days after the baseline visit (use of face masks in closed places, social distancing measures in open spaces and frequent handwashing).
7. Have been vaccinated with any of the approved vaccines against SARS-CoV-2 (at least once).

Exclusion Criteria:

1. History of hypersensibility or allergy to any of the vaccine compounds.
2. History of severe anaphylactic reactions of any cause.
3. Fever at the baseline visit.
4. Active participation in any other clinical trial or experimental intervention within last 3 months.
5. Have received any vaccine (experimental or approved) within 30 days before baseline visit, except for influenza vaccine.
6. The last anti-COVID vaccination was less than 4 months ago.
7. SARS-CoV-2 infection occurred in less than 1 month ago.
8. Pregnant or nursing women.
9. Child-bearing potential and sexually active women who do not use highly effective birth control methods (oral contraceptives, intrauterine device, subcutaneous implant, transdermal patch used at least within 3 months) at the time of enrolment. Fertile and sexually active men not willing to strictly use (in all relationships) barrier methods of birth control throughout study. Those participants (both sexes) not sexually active can participate in the study if they are committed to avoid sexual intercourse throughout study (6 months).
10. Chronic diseases that require use of immunosuppressive agents or immune response modulators (for instance: systemic corticosteroids, cyclosporine, rituximab, among others).
11. Cancer under active chemotherapy treatment.
12. Subjects with HIV infection history.
13. Subjects with chronic renal or liver disease who have shown an infectious condition that required hospitalization or treatment with intravenous drugs within the last year prior baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4065 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Phase II - Increase in titres of neutralizing anti SARS-CoV-2 IgG antibodies in serum | 14 to 17 days after vaccination
  Serum IgG, neutralizing antibodies
Phase II - T-cell elicited responses | Day 14
  Percentage of cells expressing IL2, TNF-alpha and IFN-gamma by Flow cytometry after challenge with spike protein.
Phase III - Increase in titres of neutralizing anti SARS-CoV-2 IgG antibodies in serum | 14 to 17 days after vaccination
  Serum IgG, neutralizing antibodies

SECONDARY OUTCOMES:
Phase II - Increase in titres of neutralizing anti SARS-CoV-2 IgG antibodies in serum | Day 0 (day of vaccination)
  Serum IgG, neutralizing antibodies
Phase II - Increase in titres of neutralizing anti SARS-CoV-2 IgG antibodies in serum | Day 90 after vaccination
  Serum IgG, neutralizing antibodies
Phase II - Increase in titres of neutralizing anti SARS-CoV-2 IgG antibodies in serum | Day 180 after vaccination
  Serum IgG, neutralizing antibodies
Phase II - T-cell elicited responses | Day 0 (day of vaccination)
  Percentage of cells expressing IL2, TNF-alpha and IFN-gamma by Flow cytometry after challenge with spike protein.
Phase II - T-cell elicited responses | Day 90 after vaccination
  Percentage of cells expressing IL2, TNF-alpha and IFN-gamma by Flow cytometry after challenge with spike protein.
Phase II - T-cell elicited responses | Day 180 after vaccination
  Percentage of cells expressing IL2, TNF-alpha and IFN-gamma by Flow cytometry after challenge with spike protein.
Phase III - Incidence of symptomatic COVID-19 disease cases | From 14 days after vaccination
  Document the incidence of COVID-19 disease symptomatic cases in both groups (experimental vaccine and active control).
Phase III - Incidence of severe COVID-19 disease cases or mortality | From 14 days after vaccination
  Document the incidence of severe or mortality COVID-19 disease cases in both groups (experimental vaccine and active control).

OTHER OUTCOMES:
Phase II/Phase III - Safety: Adverse Events | After Day 14 after vaccination
  Incidence of adverse events
Phase II -Basal titers of Anti-N and anti-S antibodies, distribution of anti-N and anti-S antibodies within study population | Day 0 (day of vaccination)
  Appearance of anti-N and anti-S antibodies
Phase II - Increase in titers of Anti-N and anti-S antibodies, distribution of anti-N and anti-S antibodies within study population | Day 14 after vaccination
  Appearance of anti-N and anti-S antibodies
Phase II - Increase in titers of Anti-N and anti-S antibodies, distribution of anti-N and anti-S antibodies within study population | Day 90 after vaccination
  Appearance of anti-N and anti-S antibodies
Phase II - Increase in titers of Anti-N and anti-S antibodies, distribution of anti-N and anti-S antibodies within study population | Day 180 after vaccination
  Appearance of anti-N and anti-S antibodies
Phase II - Incidence of confirmed cases of SARS-CoV-2 infection | Day 28 until the end of the study.
  Evaluation of the incidence of confirmed cases of SARS-CoV-2 infection in study subjects from systematic vaccination.
Increase in titres of neutralizing anti SARS-CoV-2 IgG antibodies in serum in selected subpopulations | From 14 and up to 180 days after vaccination
  Subjects younger than 65 years. Subjects older than 65 years. Subjects with at least one comorbidity (any). Subjects with obesity (BMI >30). Subjects with Diabetes Mellitus. Subjects with hypertension. Subjects with smoking history. Subjects with asthma.
  Subjects with cardiovascular disease. Subjects with chronic obstructive pulmonary disease. Subjects with chronic renal disease. Subjects with liver disease. Subjects with cancer history.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Peralta, Study Director — Laboratorio Avi-Mex, S.A. de C.V.
Locations (14):
- Mexico (14):
  - Promotora Médica Aguascalientes, S.A. de C.V., Aguascalientes, Aguascalientes
  - Centro de Investigación Clínica del Pacífico, S.A. de C.V., Acapulco de Juárez, Guerrero
  - Centro de Investigación Clínica Chapultepec S.A. de C.V., Coyoacán, Mexico City
  - Centro de Investigación Clínica Acelerada, S.C., Gustavo Adolfo Madero, Mexico City
  - Unidad de Medicina Familiar No. 20 - IMSS, Gustavo Adolfo Madero, Mexico City
  - CAIMED Investigación en Salud S.A. de C.V., Mexico City, Mexico City
  - Sociedad Administradora de Servicios de Salud, S.C., Morelia, Michoacán
  - Oaxaca Site Management Organization, S.C., Oaxaca City, Oaxaca
  - Centro de Investigación y Avances Médicos Especializados / RED OSMO Cancún, Cancún, Quintana Roo
  - Clinical Research Institute S.C., Tlalnepantla, State of Mexico
  - Profesionales Médicos Desarrollados, S.C. (Instituto Veracruzano de Investigación Clínica), Veracruz, Veracruz
  - Centro Multidisciplinario para el Desarrollo Especializado de la Investigación Clinica en Yucatán S.C.P., Mérida, Yucatán
  - Jules Bordet Medical Service, S.C.P. / Khöler & Milstein Research, Mérida, Yucatán
  - Unidad de Atención Médica e Investigación en Salud, S.C.P., Mérida, Yucatán

IPD SHARING:
Plan to Share IPD: Yes
Individual deidentified participant data (including data dictionaries) will not be shared, but only to the extent permitted in the informed consent and under Mexican law.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available immediately following publication and for 12 months thereafter.
Access Criteria: Data will be available only to investigators whose proposed use of the data has been authorized by an independent review committee and the ethics committees involved in the authorization of the protocol, and/or the Federal Commission for the Protection against Sanitary Risks (COFEPRIS) in Mexico if required by law. The permitted use of the data will be as authorized. Proposals or requests should be directed to gustavo.peralta@avimex.com.mx and authorized data requestors must sign a data access agreement.

REFERENCES:
- [Background] 1. Ponce de León, S. et. al. (2022) Safety and immunogenicity of a live recombinant Newcastle disease virus-based COVID-19 vaccine (Patria) administered via the intramuscular or intranasal route: Interim results of a non-randomized open label phase I trial in Mexico. Pre-Print. https://www.medrxiv.org/content/10.1101/2022.02.08.22270676v1 doi: https://doi.org/10.1101/2022.02.08.22270676
- [Background] Lara-Puente JH, Carreno JM, Sun W, Suarez-Martinez A, Ramirez-Martinez L, Quezada-Monroy F, Paz-De la Rosa G, Vigueras-Moreno R, Singh G, Rojas-Martinez O, Chagoya-Cortes HE, Sarfati-Mizrahi D, Soto-Priante E, Lopez-Macias C, Krammer F, Castro-Peralta F, Palese P, Garcia-Sastre A, Lozano-Dubernard B. Safety and Immunogenicity of a Newcastle Disease Virus Vector-Based SARS-CoV-2 Vaccine Candidate, AVX/COVID-12-HEXAPRO (Patria), in Pigs. mBio. 2021 Oct 26;12(5):e0190821. doi: 10.1128/mBio.01908-21. Epub 2021 Sep 21. PMID 34544278
- [Background] Logunov DY, Dolzhikova IV, Zubkova OV, Tukhvatullin AI, Shcheblyakov DV, Dzharullaeva AS, Grousova DM, Erokhova AS, Kovyrshina AV, Botikov AG, Izhaeva FM, Popova O, Ozharovskaya TA, Esmagambetov IB, Favorskaya IA, Zrelkin DI, Voronina DV, Shcherbinin DN, Semikhin AS, Simakova YV, Tokarskaya EA, Lubenets NL, Egorova DA, Shmarov MM, Nikitenko NA, Morozova LF, Smolyarchuk EA, Kryukov EV, Babira VF, Borisevich SV, Naroditsky BS, Gintsburg AL. Safety and immunogenicity of an rAd26 and rAd5 vector-based heterologous prime-boost COVID-19 vaccine in two formulations: two open, non-randomised phase 1/2 studies from Russia. Lancet. 2020 Sep 26;396(10255):887-897. doi: 10.1016/S0140-6736(20)31866-3. Epub 2020 Sep 4. PMID 32896291
- [Background] Determining Sample Sizes Needed to Detect a Difference between Two Proportions. In: Statistical Methods for Rates and Proportions. John Wiley & Sons, Ltd, 2003: 64-85.
- [Background] Ritchie H, Ortiz-Ospina E, Beltekian D, et al. Coronavirus Pandemic (COVID-19). Our World in Data 2020; published online March 5. https://ourworldindata.org/covid-cases (accessed Aug 2, 2021).
- [Background] Exceso de Mortalidad en México - Coronavirus. https://coronavirus.gob.mx/exceso-de-mortalidad-en-mexico/ (accessed Aug 2, 2021).
- [Background] Dhillon P, Altmann D, Male V. COVID-19 vaccines: what do we know so far? FEBS J. 2021 Sep;288(17):4996-5009. doi: 10.1111/febs.16094. Epub 2021 Jul 19. PMID 34288409
- [Background] Zamai L, Rocchi MBL. Hypothesis: Possible influence of antivector immunity and SARS-CoV-2 variants on efficacy of ChAdOx1 nCoV-19 vaccine. Br J Pharmacol. 2022 Jan;179(2):218-226. doi: 10.1111/bph.15620. Epub 2021 Jul 31. PMID 34331459
- [Background] Barros-Martins J, Hammerschmidt SI, Cossmann A, Odak I, Stankov MV, Morillas Ramos G, Dopfer-Jablonka A, Heidemann A, Ritter C, Friedrichsen M, Schultze-Florey C, Ravens I, Willenzon S, Bubke A, Ristenpart J, Janssen A, Ssebyatika G, Bernhardt G, Munch J, Hoffmann M, Pohlmann S, Krey T, Bosnjak B, Forster R, Behrens GMN. Immune responses against SARS-CoV-2 variants after heterologous and homologous ChAdOx1 nCoV-19/BNT162b2 vaccination. Nat Med. 2021 Sep;27(9):1525-1529. doi: 10.1038/s41591-021-01449-9. Epub 2021 Jul 14. PMID 34262158
- [Background] He Q, Mao Q, An C, Zhang J, Gao F, Bian L, Li C, Liang Z, Xu M, Wang J. Heterologous prime-boost: breaking the protective immune response bottleneck of COVID-19 vaccine candidates. Emerg Microbes Infect. 2021 Dec;10(1):629-637. doi: 10.1080/22221751.2021.1902245. PMID 33691606
- [Background] Normark J, Vikstrom L, Gwon YD, Persson IL, Edin A, Bjorsell T, Dernstedt A, Christ W, Tevell S, Evander M, Klingstrom J, Ahlm C, Forsell M. Heterologous ChAdOx1 nCoV-19 and mRNA-1273 Vaccination. N Engl J Med. 2021 Sep 9;385(11):1049-1051. doi: 10.1056/NEJMc2110716. Epub 2021 Jul 14. No abstract available. PMID 34260850
- [Background] Hill JA, Ujjani CS, Greninger AL, Shadman M, Gopal AK. Immunogenicity of a heterologous COVID-19 vaccine after failed vaccination in a lymphoma patient. Cancer Cell. 2021 Aug 9;39(8):1037-1038. doi: 10.1016/j.ccell.2021.06.015. Epub 2021 Jun 26. No abstract available. PMID 34242571
- [Background] Velasco M, Galan MI, Casas ML, Perez-Fernandez E, Martinez-Ponce D, Gonzalez-Pineiro B, Castilla V, Guijarro C; Alcorcon COVID-19 Working Group. Impact of Previous Coronavirus Disease 2019 on Immune Response After a Single Dose of BNT162b2 Severe Acute Respiratory Syndrome Coronavirus 2 Vaccine. Open Forum Infect Dis. 2021 Jun 4;8(7):ofab299. doi: 10.1093/ofid/ofab299. eCollection 2021 Jul. PMID 34258322
- [Background] Levi R, Azzolini E, Pozzi C, Ubaldi L, Lagioia M, Mantovani A, Rescigno M. One dose of SARS-CoV-2 vaccine exponentially increases antibodies in individuals who have recovered from symptomatic COVID-19. J Clin Invest. 2021 Jun 15;131(12):e149154. doi: 10.1172/JCI149154. PMID 33956667
- [Background] Reynolds CJ, Pade C, Gibbons JM, Butler DK, Otter AD, Menacho K, Fontana M, Smit A, Sackville-West JE, Cutino-Moguel T, Maini MK, Chain B, Noursadeghi M; UK COVIDsortium Immune Correlates Network; Brooks T, Semper A, Manisty C, Treibel TA, Moon JC; UK COVIDsortium Investigators; Valdes AM, McKnight A, Altmann DM, Boyton R. Prior SARS-CoV-2 infection rescues B and T cell responses to variants after first vaccine dose. Science. 2021 Apr 30;372(6549):1418-23. doi: 10.1126/science.abh1282. Online ahead of print. PMID 33931567
- [Background] Commissioner O of the. Joint Statement from HHS Public Health and Medical Experts on COVID-19 Booster Shots. FDA. 2021; published online Aug 18. https://www.fda.gov/news-events/press-announcements/joint-statement-hhs-public-health-and-medical-experts-covid-19-booster-shots (accessed Aug 19, 2021).
- [Background] Sun W, Leist SR, McCroskery S, Liu Y, Slamanig S, Oliva J, Amanat F, Schafer A, Dinnon KH 3rd, Garcia-Sastre A, Krammer F, Baric RS, Palese P. Newcastle disease virus (NDV) expressing the spike protein of SARS-CoV-2 as a live virus vaccine candidate. EBioMedicine. 2020 Dec;62:103132. doi: 10.1016/j.ebiom.2020.103132. Epub 2020 Nov 21. PMID 33232870
- [Background] DiNapoli JM, Kotelkin A, Yang L, Elankumaran S, Murphy BR, Samal SK, Collins PL, Bukreyev A. Newcastle disease virus, a host range-restricted virus, as a vaccine vector for intranasal immunization against emerging pathogens. Proc Natl Acad Sci U S A. 2007 Jun 5;104(23):9788-93. doi: 10.1073/pnas.0703584104. Epub 2007 May 29. PMID 17535926
- [Background] Bukreyev A, Huang Z, Yang L, Elankumaran S, St Claire M, Murphy BR, Samal SK, Collins PL. Recombinant newcastle disease virus expressing a foreign viral antigen is attenuated and highly immunogenic in primates. J Virol. 2005 Nov;79(21):13275-84. doi: 10.1128/JVI.79.21.13275-13284.2005. PMID 16227250
- [Background] Brown CM, Vostok J, Johnson H, Burns M, Gharpure R, Sami S, Sabo RT, Hall N, Foreman A, Schubert PL, Gallagher GR, Fink T, Madoff LC, Gabriel SB, MacInnis B, Park DJ, Siddle KJ, Harik V, Arvidson D, Brock-Fisher T, Dunn M, Kearns A, Laney AS. Outbreak of SARS-CoV-2 Infections, Including COVID-19 Vaccine Breakthrough Infections, Associated with Large Public Gatherings - Barnstable County, Massachusetts, July 2021. MMWR Morb Mortal Wkly Rep. 2021 Aug 6;70(31):1059-1062. doi: 10.15585/mmwr.mm7031e2. PMID 34351882
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Chan JF, Yuan S, Kok KH, To KK, Chu H, Yang J, Xing F, Liu J, Yip CC, Poon RW, Tsoi HW, Lo SK, Chan KH, Poon VK, Chan WM, Ip JD, Cai JP, Cheng VC, Chen H, Hui CK, Yuen KY. A familial cluster of pneumonia associated with the 2019 novel coronavirus indicating person-to-person transmission: a study of a family cluster. Lancet. 2020 Feb 15;395(10223):514-523. doi: 10.1016/S0140-6736(20)30154-9. Epub 2020 Jan 24. PMID 31986261
- [Background] Chan JF, Kok KH, Zhu Z, Chu H, To KK, Yuan S, Yuen KY. Genomic characterization of the 2019 novel human-pathogenic coronavirus isolated from a patient with atypical pneumonia after visiting Wuhan. Emerg Microbes Infect. 2020 Jan 28;9(1):221-236. doi: 10.1080/22221751.2020.1719902. eCollection 2020. PMID 31987001
- [Background] Wu F, Zhao S, Yu B, Chen YM, Wang W, Song ZG, Hu Y, Tao ZW, Tian JH, Pei YY, Yuan ML, Zhang YL, Dai FH, Liu Y, Wang QM, Zheng JJ, Xu L, Holmes EC, Zhang YZ. A new coronavirus associated with human respiratory disease in China. Nature. 2020 Mar;579(7798):265-269. doi: 10.1038/s41586-020-2008-3. Epub 2020 Feb 3. PMID 32015508
- [Background] Wan Y, Shang J, Graham R, Baric RS, Li F. Receptor Recognition by the Novel Coronavirus from Wuhan: an Analysis Based on Decade-Long Structural Studies of SARS Coronavirus. J Virol. 2020 Mar 17;94(7):e00127-20. doi: 10.1128/JVI.00127-20. Print 2020 Mar 17. PMID 31996437
- [Background] Hoffmann M, Kleine-Weber H, Schroeder S, Kruger N, Herrler T, Erichsen S, Schiergens TS, Herrler G, Wu NH, Nitsche A, Muller MA, Drosten C, Pohlmann S. SARS-CoV-2 Cell Entry Depends on ACE2 and TMPRSS2 and Is Blocked by a Clinically Proven Protease Inhibitor. Cell. 2020 Apr 16;181(2):271-280.e8. doi: 10.1016/j.cell.2020.02.052. Epub 2020 Mar 5. PMID 32142651
- [Background] Yao H, Song Y, Chen Y, Wu N, Xu J, Sun C, Zhang J, Weng T, Zhang Z, Wu Z, Cheng L, Shi D, Lu X, Lei J, Crispin M, Shi Y, Li L, Li S. Molecular Architecture of the SARS-CoV-2 Virus. Cell. 2020 Oct 29;183(3):730-738.e13. doi: 10.1016/j.cell.2020.09.018. Epub 2020 Sep 6. PMID 32979942
- [Background] Wrapp D, Wang N, Corbett KS, Goldsmith JA, Hsieh CL, Abiona O, Graham BS, McLellan JS. Cryo-EM structure of the 2019-nCoV spike in the prefusion conformation. Science. 2020 Mar 13;367(6483):1260-1263. doi: 10.1126/science.abb2507. Epub 2020 Feb 19. PMID 32075877
- [Background] Piccoli L, Park YJ, Tortorici MA, Czudnochowski N, Walls AC, Beltramello M, Silacci-Fregni C, Pinto D, Rosen LE, Bowen JE, Acton OJ, Jaconi S, Guarino B, Minola A, Zatta F, Sprugasci N, Bassi J, Peter A, De Marco A, Nix JC, Mele F, Jovic S, Rodriguez BF, Gupta SV, Jin F, Piumatti G, Lo Presti G, Pellanda AF, Biggiogero M, Tarkowski M, Pizzuto MS, Cameroni E, Havenar-Daughton C, Smithey M, Hong D, Lepori V, Albanese E, Ceschi A, Bernasconi E, Elzi L, Ferrari P, Garzoni C, Riva A, Snell G, Sallusto F, Fink K, Virgin HW, Lanzavecchia A, Corti D, Veesler D. Mapping Neutralizing and Immunodominant Sites on the SARS-CoV-2 Spike Receptor-Binding Domain by Structure-Guided High-Resolution Serology. Cell. 2020 Nov 12;183(4):1024-1042.e21. doi: 10.1016/j.cell.2020.09.037. Epub 2020 Sep 16. PMID 32991844
- [Background] Tan CW, Chia WN, Qin X, Liu P, Chen MI, Tiu C, Hu Z, Chen VC, Young BE, Sia WR, Tan YJ, Foo R, Yi Y, Lye DC, Anderson DE, Wang LF. A SARS-CoV-2 surrogate virus neutralization test based on antibody-mediated blockage of ACE2-spike protein-protein interaction. Nat Biotechnol. 2020 Sep;38(9):1073-1078. doi: 10.1038/s41587-020-0631-z. Epub 2020 Jul 23. PMID 32704169
- [Background] Chen X, Pan Z, Yue S, Yu F, Zhang J, Yang Y, Li R, Liu B, Yang X, Gao L, Li Z, Lin Y, Huang Q, Xu L, Tang J, Hu L, Zhao J, Liu P, Zhang G, Chen Y, Deng K, Ye L. Disease severity dictates SARS-CoV-2-specific neutralizing antibody responses in COVID-19. Signal Transduct Target Ther. 2020 Sep 2;5(1):180. doi: 10.1038/s41392-020-00301-9. PMID 32879307
- [Background] Liu L, To KK, Chan KH, Wong YC, Zhou R, Kwan KY, Fong CH, Chen LL, Choi CY, Lu L, Tsang OT, Leung WS, To WK, Hung IF, Yuen KY, Chen Z. High neutralizing antibody titer in intensive care unit patients with COVID-19. Emerg Microbes Infect. 2020 Dec;9(1):1664-1670. doi: 10.1080/22221751.2020.1791738. PMID 32618497
- [Background] Choe PG, Kang CK, Suh HJ, Jung J, Kang E, Lee SY, Song KH, Kim HB, Kim NJ, Park WB, Kim ES, Oh MD. Antibody Responses to SARS-CoV-2 at 8 Weeks Postinfection in Asymptomatic Patients. Emerg Infect Dis. 2020 Oct;26(10):2484-2487. doi: 10.3201/eid2610.202211. Epub 2020 Jun 24. PMID 32579877
- [Background] Le Bert N, Tan AT, Kunasegaran K, Tham CYL, Hafezi M, Chia A, Chng MHY, Lin M, Tan N, Linster M, Chia WN, Chen MI, Wang LF, Ooi EE, Kalimuddin S, Tambyah PA, Low JG, Tan YJ, Bertoletti A. SARS-CoV-2-specific T cell immunity in cases of COVID-19 and SARS, and uninfected controls. Nature. 2020 Aug;584(7821):457-462. doi: 10.1038/s41586-020-2550-z. Epub 2020 Jul 15. PMID 32668444
- [Background] Dessie ZG, Zewotir T. Mortality-related risk factors of COVID-19: a systematic review and meta-analysis of 42 studies and 423,117 patients. BMC Infect Dis. 2021 Aug 21;21(1):855. doi: 10.1186/s12879-021-06536-3. PMID 34418980
- [Background] Wang Y, Perlman S. COVID-19: Inflammatory Profile. Annu Rev Med. 2022 Jan 27;73:65-80. doi: 10.1146/annurev-med-042220-012417. Epub 2021 Aug 26. PMID 34437814
- [Background] Wagner C, Griesel M, Mikolajewska A, Mueller A, Nothacker M, Kley K, Metzendorf MI, Fischer AL, Kopp M, Stegemann M, Skoetz N, Fichtner F. Systemic corticosteroids for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Aug 16;8(8):CD014963. doi: 10.1002/14651858.CD014963. PMID 34396514
- [Background] Ansems K, Grundeis F, Dahms K, Mikolajewska A, Thieme V, Piechotta V, Metzendorf MI, Stegemann M, Benstoem C, Fichtner F. Remdesivir for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD014962. doi: 10.1002/14651858.CD014962. PMID 34350582
- [Background] Ghosn L, Chaimani A, Evrenoglou T, Davidson M, Grana C, Schmucker C, Bollig C, Henschke N, Sguassero Y, Nejstgaard CH, Menon S, Nguyen TV, Ferrand G, Kapp P, Riveros C, Avila C, Devane D, Meerpohl JJ, Rada G, Hrobjartsson A, Grasselli G, Tovey D, Ravaud P, Boutron I. Interleukin-6 blocking agents for treating COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 Mar 18;3(3):CD013881. doi: 10.1002/14651858.CD013881. PMID 33734435
- [Background] Khoury DS, Cromer D, Reynaldi A, Schlub TE, Wheatley AK, Juno JA, Subbarao K, Kent SJ, Triccas JA, Davenport MP. Neutralizing antibody levels are highly predictive of immune protection from symptomatic SARS-CoV-2 infection. Nat Med. 2021 Jul;27(7):1205-1211. doi: 10.1038/s41591-021-01377-8. Epub 2021 May 17. PMID 34002089
- [Background] Liu A, Li Y, Peng J, Huang Y, Xu D. Antibody responses against SARS-CoV-2 in COVID-19 patients. J Med Virol. 2021 Jan;93(1):144-148. doi: 10.1002/jmv.26241. Epub 2020 Aug 2. No abstract available. PMID 32603501
- [Background] Perreault J, Tremblay T, Fournier MJ, Drouin M, Beaudoin-Bussieres G, Prevost J, Lewin A, Begin P, Finzi A, Bazin R. Waning of SARS-CoV-2 RBD antibodies in longitudinal convalescent plasma samples within 4 months after symptom onset. Blood. 2020 Nov 26;136(22):2588-2591. doi: 10.1182/blood.2020008367. PMID 33001206
- [Background] Post N, Eddy D, Huntley C, van Schalkwyk MCI, Shrotri M, Leeman D, Rigby S, Williams SV, Bermingham WH, Kellam P, Maher J, Shields AM, Amirthalingam G, Peacock SJ, Ismail SA. Antibody response to SARS-CoV-2 infection in humans: A systematic review. PLoS One. 2020 Dec 31;15(12):e0244126. doi: 10.1371/journal.pone.0244126. eCollection 2020. PMID 33382764
- [Background] Juthani PV, Gupta A, Borges KA, Price CC, Lee AI, Won CH, Chun HJ. Hospitalisation among vaccine breakthrough COVID-19 infections. Lancet Infect Dis. 2021 Nov;21(11):1485-1486. doi: 10.1016/S1473-3099(21)00558-2. Epub 2021 Sep 7. No abstract available. PMID 34506735
- [Background] Borobia AM, Carcas AJ, Perez-Olmeda M, Castano L, Bertran MJ, Garcia-Perez J, Campins M, Portoles A, Gonzalez-Perez M, Garcia Morales MT, Arana-Arri E, Aldea M, Diez-Fuertes F, Fuentes I, Ascaso A, Lora D, Imaz-Ayo N, Baron-Mira LE, Agusti A, Perez-Ingidua C, Gomez de la Camara A, Arribas JR, Ochando J, Alcami J, Belda-Iniesta C, Frias J; CombiVacS Study Group. Immunogenicity and reactogenicity of BNT162b2 booster in ChAdOx1-S-primed participants (CombiVacS): a multicentre, open-label, randomised, controlled, phase 2 trial. Lancet. 2021 Jul 10;398(10295):121-130. doi: 10.1016/S0140-6736(21)01420-3. Epub 2021 Jun 25. PMID 34181880
- [Background] Hsieh CL, Goldsmith JA, Schaub JM, DiVenere AM, Kuo HC, Javanmardi K, Le KC, Wrapp D, Lee AG, Liu Y, Chou CW, Byrne PO, Hjorth CK, Johnson NV, Ludes-Meyers J, Nguyen AW, Park J, Wang N, Amengor D, Lavinder JJ, Ippolito GC, Maynard JA, Finkelstein IJ, McLellan JS. Structure-based design of prefusion-stabilized SARS-CoV-2 spikes. Science. 2020 Sep 18;369(6510):1501-1505. doi: 10.1126/science.abd0826. Epub 2020 Jul 23. PMID 32703906
- [Background] Rodda LB, Netland J, Shehata L, Pruner KB, Morawski PA, Thouvenel CD, Takehara KK, Eggenberger J, Hemann EA, Waterman HR, Fahning ML, Chen Y, Hale M, Rathe J, Stokes C, Wrenn S, Fiala B, Carter L, Hamerman JA, King NP, Gale M Jr, Campbell DJ, Rawlings DJ, Pepper M. Functional SARS-CoV-2-Specific Immune Memory Persists after Mild COVID-19. Cell. 2021 Jan 7;184(1):169-183.e17. doi: 10.1016/j.cell.2020.11.029. Epub 2020 Nov 23. PMID 33296701
- [Background] Barouch DH, Stephenson KE, Sadoff J, Yu J, Chang A, Gebre M, McMahan K, Liu J, Chandrashekar A, Patel S, Le Gars M, de Groot AM, Heerwegh D, Struyf F, Douoguih M, van Hoof J, Schuitemaker H. Durable Humoral and Cellular Immune Responses 8 Months after Ad26.COV2.S Vaccination. N Engl J Med. 2021 Sep 2;385(10):951-953. doi: 10.1056/NEJMc2108829. Epub 2021 Jul 14. No abstract available. PMID 34260834
- [Background] Thomas SJ, Moreira ED Jr, Kitchin N, Absalon J, Gurtman A, Lockhart S, Perez JL, Perez Marc G, Polack FP, Zerbini C, Bailey R, Swanson KA, Xu X, Roychoudhury S, Koury K, Bouguermouh S, Kalina WV, Cooper D, Frenck RW Jr, Hammitt LL, Tureci O, Nell H, Schaefer A, Unal S, Yang Q, Liberator P, Tresnan DB, Mather S, Dormitzer PR, Sahin U, Gruber WC, Jansen KU; C4591001 Clinical Trial Group. Safety and Efficacy of the BNT162b2 mRNA Covid-19 Vaccine through 6 Months. N Engl J Med. 2021 Nov 4;385(19):1761-1773. doi: 10.1056/NEJMoa2110345. Epub 2021 Sep 15. PMID 34525277
- [Background] Lopez Bernal J, Andrews N, Gower C, Gallagher E, Simmons R, Thelwall S, Stowe J, Tessier E, Groves N, Dabrera G, Myers R, Campbell CNJ, Amirthalingam G, Edmunds M, Zambon M, Brown KE, Hopkins S, Chand M, Ramsay M. Effectiveness of Covid-19 Vaccines against the B.1.617.2 (Delta) Variant. N Engl J Med. 2021 Aug 12;385(7):585-594. doi: 10.1056/NEJMoa2108891. Epub 2021 Jul 21. PMID 34289274
- [Background] Hacisuleyman E, Hale C, Saito Y, Blachere NE, Bergh M, Conlon EG, Schaefer-Babajew DJ, DaSilva J, Muecksch F, Gaebler C, Lifton R, Nussenzweig MC, Hatziioannou T, Bieniasz PD, Darnell RB. Vaccine Breakthrough Infections with SARS-CoV-2 Variants. N Engl J Med. 2021 Jun 10;384(23):2212-2218. doi: 10.1056/NEJMoa2105000. Epub 2021 Apr 21. PMID 33882219
- [Background] Bergwerk M, Gonen T, Lustig Y, Amit S, Lipsitch M, Cohen C, Mandelboim M, Levin EG, Rubin C, Indenbaum V, Tal I, Zavitan M, Zuckerman N, Bar-Chaim A, Kreiss Y, Regev-Yochay G. Covid-19 Breakthrough Infections in Vaccinated Health Care Workers. N Engl J Med. 2021 Oct 14;385(16):1474-1484. doi: 10.1056/NEJMoa2109072. Epub 2021 Jul 28. PMID 34320281
- [Background] Keehner J, Horton LE, Binkin NJ, Laurent LC; SEARCH Alliance; Pride D, Longhurst CA, Abeles SR, Torriani FJ. Resurgence of SARS-CoV-2 Infection in a Highly Vaccinated Health System Workforce. N Engl J Med. 2021 Sep 30;385(14):1330-1332. doi: 10.1056/NEJMc2112981. Epub 2021 Sep 1. No abstract available. PMID 34469645
- [Background] Mathieu E, Ritchie H, Ortiz-Ospina E, Roser M, Hasell J, Appel C, Giattino C, Rodes-Guirao L. A global database of COVID-19 vaccinations. Nat Hum Behav. 2021 Jul;5(7):947-953. doi: 10.1038/s41562-021-01122-8. Epub 2021 May 10. PMID 33972767
- [Background] Macpherson LW. Some Observations On The Epizootiology Of NewCastle Disease. Can J Comp Med Vet Sci. 1956 May;20(5):155-68. No abstract available. PMID 17648892
- [Background] Alexander DJ. Newcastle disease and other avian paramyxoviruses. Rev Sci Tech. 2000 Aug;19(2):443-62. doi: 10.20506/rst.19.2.1231. PMID 10935273
- [Background] NELSON CB, POMEROY BS, SCHRALL K, PARK WE, LINDEMAN RJ. An outbreak of conjunctivitis due to Newcastle disease virus (NDV) occurring in poultry workers. Am J Public Health Nations Health. 1952 Jun;42(6):672-8. doi: 10.2105/ajph.42.6.672. No abstract available. PMID 14924001
- [Background] Kim SH, Samal SK. Newcastle Disease Virus as a Vaccine Vector for Development of Human and Veterinary Vaccines. Viruses. 2016 Jul 4;8(7):183. doi: 10.3390/v8070183. PMID 27384578
- [Background] Sun W, McCroskery S, Liu WC, Leist SR, Liu Y, Albrecht RA, Slamanig S, Oliva J, Amanat F, Schafer A, Dinnon KH 3rd, Innis BL, Garcia-Sastre A, Krammer F, Baric RS, Palese P. A Newcastle Disease Virus (NDV) Expressing a Membrane-Anchored Spike as a Cost-Effective Inactivated SARS-CoV-2 Vaccine. Vaccines (Basel). 2020 Dec 17;8(4):771. doi: 10.3390/vaccines8040771. PMID 33348607
- [Background] Naranjo CA, Busto U, Sellers EM, Sandor P, Ruiz I, Roberts EA, Janecek E, Domecq C, Greenblatt DJ. A method for estimating the probability of adverse drug reactions. Clin Pharmacol Ther. 1981 Aug;30(2):239-45. doi: 10.1038/clpt.1981.154. No abstract available. PMID 7249508